CLINICAL TRIAL: NCT04997564
Title: The Efficacy and Safety of 12-week SOF/VEL Regimen Combined With Prophylactic Use of TAF for Treatment-naïve Genotype 1-6 HCV/HBV Co-infection Adult Patients With or Without Compensated Cirrhosis in China : a Mutil-center,Prospective,Single-arm,Open-label Trial
Brief Title: The Efficacy and Safety of 12-week SOF/VEL Regimen Combined With Prophylactic Use of TAF for Treatment-naïve Genotype 1-6 HCV/HBV Co-infection Adult Patients With or Without Compensated Cirrhosis in China
Acronym: BDTAF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Xiaoyuan XU, professor, Peking University First Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021XXYU-study
Record Dates: First submitted 2021-07-13; First posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Chronic Hepatitis C; Chronic Hepatitis B
Keywords: chronic hepatitis B virus (HBV); hepatitis C virus (HCV)
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis B, Chronic; Hepatitis C | interventions — tenofovir alafenamide; sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-cirrhotic patients (Experimental): patients will be discontinued TAF once daily therapy at the end of week 28 if no HBV reactivation occurs during treatment
  Interventions: Drug: Tenofovir Alafenamide 25 MG; Drug: Sofosbuvir / Velpatasvir
- cirrhotic patients (Other): patients will be received TAF once daily for 64 weeks. In this study, after week 64, and patients will continue NUC treatment but pay by themselves.
  Interventions: Drug: Tenofovir Alafenamide 25 MG; Drug: Sofosbuvir / Velpatasvir

INTERVENTIONS:
Drug: Tenofovir Alafenamide 25 MG — All the patients will use prophylactically TAF for 4 weeks before using SOF/VEL once daily for 12 weeks. Group 1 patients will be discontinued TAF once daily therapy at the end of week 28 if no HBV reactivation occurs during treatment .
Drug: Sofosbuvir / Velpatasvir — All the patients will use prophylactically TAF for 4 weeks before using SOF/VEL once daily for 12 weeks. Group 2 patients will be received TAF once daily for 64 weeks. In this study, after week 64.

SUMMARY:
Subjects can be classified into two groups, Group 1 include non-cirrhotic patients, Group 2 include cirrhotic patients.

All the patients will be received prophylactically TAF for 4 weeks before using SOF/VEL once daily for 12 weeks. In total, Group 1 patients will be discontinued TAF once daily therapy at the end of week 28 if no HBV reactivation occurs during treatment , Group 2 patients will be received TAF once daily for 64 weeks. In this study, after week 64, Group 2 patients will continue NUC treatment but pay by themselves. For those who is GT3 cirrhosis patients, RBV added simultaneously with SOF/VEL for 12 weeks. For patients weighing < 75 kg, the dose is 500 mg twice; for patients weighing ≥ 75 kg, the dose is 600 mg twice.

DETAILED DESCRIPTION:
Subjects can be classified into two groups, Group 1 include non-cirrhotic patients, Group 2 include cirrhotic patients.

All the patients will be received prophylactically TAF for 4 weeks before using SOF/VEL once daily for 12 weeks. In total, Group 1 patients will be discontinued TAF once daily therapy at the end of week 28 if no HBV reactivation occurs during treatment , Group 2 patients will be received TAF once daily for 64 weeks. In this study, after week 64, Group 2 patients will continue NUC treatment but pay by themselves. For those who is GT3 cirrhosis patients, RBV added simultaneously with SOF/VEL for 12 weeks. For patients weighing < 75 kg, the dose is 500 mg twice; for patients weighing ≥ 75 kg, the dose is 600 mg twice.

The primary objective of this study is:

•To evaluate efficacy and safety of SOF/VEL in HBsAg-positive patients with HCV (GT1-6) co-infection.

The secondary objectives of this study are:

* To evaluate the proportion of subjects with HBV reactivation during the treatment and after cessation of treatment.
* To evaluate the proportion of subjects with virologic failure (virological breakthrough/ viral relapse)of HCV/ HBV.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent
2. Male or female, age≥18 years
3. Bodyweight≥40 kg
4. HCV RNA positive (15 IU/mL )at Screening
5. HCV genotype 1, 2, 3, 4, 5, 6, or indeterminate as assessed at Screening by the Central Laboratory
6. Chronic HBV/HCV coinfection (≥ 6 months) documented by prior medical history or liver biopsy. For non-cirrhotic patients, and for HBeAg positive patients, HBV DNA<20000IU/ml. For HBeAg negative patients, HBV DNA<2000IU/ml.

   For cirrhosis patients, HBV DNA was dectable or undectable. Cirrhosis Determination (approximately 20% of subjects may have cirrhosis)
   * Cirrhosis by B Ultrasound/CT/ MRI.
   * Cirrhosis is defined as Fibroscan® with a result of ≥ 17.5 kPa
   * Absence of cirrhosis is defined as Fibroscan with a result of <10.6 kPa within ≤ 6 months of Day 1
7. Classification as treatment naïve for CHC patients Treatment naïve is defined as having never been exposed to approved or experimental HCV-specific direct-acting antiviral agents or prior treatment of HCV with interferon or ribavirin
8. Individuals must not be taking or requiring treatment with HBV antiviral therapy at screening. For participants that are HBV treatment experienced, the most recent treatment must have been completed at least 6 months prior to Day 1.
9. Patients with HBsAg positive as least 6 month without decompensated cirrhosis.
10. Liver imaging within 6 months of Day 1 is required in cirrhotic patients only to exclude hepatocellular carcinoma (HCC)
11. Females of childbearing potential (as defined in Appendix 4) must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day 1 prior to enrollment
12. Male subjects and female subjects of childbearing potential who engage in heterosexualinter course must agree to use protocol specified method(s) of contraception as described in Appendix 4
13. Lactating females must agree to discontinue nursing before the study drug is administered
14. Subject must be of generally good health, with the exception of chronic HBV/HCV infection, as determined by the Investigator
15. Subject must be able to comply with the dosing instructions for study drug administration and able to complete the study -

Exclusion Criteria:

1. Any direct antiviral drugs (DAAs) used before screening, including non-structural proteins NS3/4A inhibitor, NS5A inhibitor or NS5B polymerase inhibitor.
2. Patients who received hepatitis B antiviral therapy within 6 months.
3. Diagnosis of primary liver cancer or support for the following evidence: alpha-fetoprotein (AFP) >100 ng/ml or cirrhosis imaging studies of the liver revealed suspicious nodules in the liver
4. A history of malignant tumors within 5 years prior to screening, except for specific cancers that have been cured by surgical resection (eg.Basal cell skin cancer, etc.), or patients suspected of having malignant tumors
5. Current or previous evidence of liver decompensation, including but not limited to: Child-Pugh score Grade B or C, ascites, or hepatic encephalopathy, variceal bleeding or diuretics for the treatment of ascites.
6. A current or previous history of a major medical condition or any other major medical disorder that may interfere with the individual's treatment, assessment or compliance program.

   1. Clinically significant disease (except HBV, HCV) or any other major disease that may interfere with subject treatment, assessment, or protocol compliance; subjects that are currently undergoing assessment of a potentially clinically significant disease (except HBV，HCV) are also excluded.
   2. Gastrointestinal disease, or the condition after surgery may interfere with the absorption of the study drug.
   3. Difficulty in collecting blood and/or poor venous access for blood collection.
   4. Solid organ transplantation.
   5. Severe lung disease, severe heart disease or porphyria.
   6. Psychiatric hospitalization, attempted suicide and/or a period of disability due to mental illness in the past 5 years. Subjects with psychiatric illness (without previously mentioned conditions) who are well-controlled or who have not needed medication for the past 12 months before Day 1 may Will be included in the study.
   7. Serious drug allergies (such as allergic reactions or hepatotoxicity).
7. Pregnant or lactating women.
8. HIV or HDV infection.
9. Screening ECG for clinically significant abnormalities
10. Subjects have the following laboratory test parameters at screening:

    1. ALT > 10 Upper Limit of Normal (ULN)
    2. AST > 10 ULN
    3. Direct bilirubin > 1.5 ULN
    4. platelets < 50,000/L
    5. HbA1c > 8.5%
    6. eGFR < 30 mL/min/1.73 m2，estimated glomerular filtration rate (eGFR) using the Cockcroft-Gault equation，eGFR will be calculated by the Cockcroft-Gault method: eGFRCG (mL/min) = [(140 - age (yrs))× weight (kg) × (0.85 if female)] / (serum creatinine (mg/dL) × 72), where weight is total body mass in kilograms.
    7. Female subjects with hemoglobin < 11 g/dL; male subjects with hemoglobin < 12 g/dL
    8. albumin < 3 g/dL
    9. INR > 1.5 x ULN unless the subject has known hemophilia or remains stable for anticoagulant therapy affecting INR
11. Chronic liver disease other than HCV pathogens (eg hemochromatosis, Wilson's disease, alpha-1 antitrypsin deficiency, cholangitis).
12. Known hypersensitivity to SOF/VEL, TAF and RBV (only for GT 3 cirrhosis patients).

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of treatment with SOF/VEL for 12 weeks in subjects with GT1-6 HCV/HBV co-infection as measured by the proportion of subjects with SVR. | The first group of patients was evaluated from 16 weeks to 28 weeks（for 12 weeks）
  hepatitis C virus is a chronic viral hepatitis caused by hepatitis C virus infection in the human body, it belongs to the liver virus, after the invasion of the human body, mainly into the human liver, can lead to chronic hepatitis
To evaluate the efficacy of treatment with SOF/VEL for 12 weeks in subjects with GT1-6 HCV/HBV co-infection as measured by the proportion of subjects with SVR. | The second group of patients was evaluated from 16 weeks to 28 weeks（for 12 weeks）
  hepatitis C virus is a chronic viral hepatitis caused by hepatitis C virus infection in the human body, it belongs to the liver virus, after the invasion of the human body, mainly into the human liver, can lead to chronic hepatitis

SECONDARY OUTCOMES:
To evaluate the proportion of subjects with HBV reactivation during the treatment and after cessation of treatment | From the commencement of SOF/VEL treatment(week 4) to week 64.
  The proportion of subjects with HBV is an acute and chronic liver disease caused by hepatitis B virus infection, which can be transmitted through blood, body fluids, contact, sexual contact transmission and vertical transmission of mother and child
To evaluate the proportion of subjects with virologic failure (virological breakthrough/ viral relapse)of HCV | The first group of patients was evaluated at week 16 to week 28
  The proportion of subjects with HCV is one of several viruses that cause viral hepatitis.
To evaluate the proportion of subjects with virologic failure (virological breakthrough/ viral relapse)of HCV | The second group of patients was evaluated at week 16 to week 64
  The proportion of subjects with HCV is one of several viruses that cause viral hepatitis.
To evaluate the proportion of subjects with virologic failure (virological breakthrough/ viral relapse)of HBV | The first group of patients was evaluated at week 4 to week 28
  The proportion of subjects with HBV is an acute and chronic liver disease caused by hepatitis B virus infection, which can be transmitted through blood, body fluids, contact, sexual contact transmission and vertical transmission of mother and child
To evaluate the proportion of subjects with virologic failure (virological breakthrough/ viral relapse)of HBV | The second group of patients was evaluated at week 4 to week 64
  The proportion of subjects with HBV is an acute and chronic liver disease caused by hepatitis B virus infection, which can be transmitted through blood, body fluids, contact, sexual contact transmission and vertical transmission of mother and child

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China